CLINICAL TRIAL: NCT00368134
Title: A Multicenter, Randomized, Double-Blind, Active-Controlled Study to Compare the Effects of 12 Weeks Treatment With Vildagliptin 50 mg Bid to Voglibose 0.2 mg Tid in Patients With Type 2 Diabetes
Brief Title: To Compare the Efficacy and Safey of Vildagliptin Compared to Voglibose in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A1301
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2007-06-28 (Estimated); Status verified 2007-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes; Vildagliptin; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin

SUMMARY:
This study is designed to evaluate the efficacy, safety and tolerability of vildagliptin compared to voglibose in patients with type 2 diabetes. Please note this study is not being conducted in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis as Type 2 Diabetes
* Patients who have been placed on dietary therapy/exercise therapy, without achievement of glycemic control
* Outpatients

Exclusion Criteria:

* Type 1 diabetes mellitus, diabetes that is a result of pancreatic injury, or secondary forms of diabetes
* Significant heart diseases
* Significant diabetic complications

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 370
Dates: Start 2006-08

PRIMARY OUTCOMES:
Change in HbA1c after 12 weeks

SECONDARY OUTCOMES:
Change in FPG after 12 weeks
Change in Fasting Lipids after 12 weeks
Change in HOMA-IR after 12 weeks
Change in HOMA-B after 12 weeks
Safety Profile after 12 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Tokyo, Japan